CLINICAL TRIAL: NCT01727466
Title: A Randomized Trial: Group Cognitive Behavior Therapy for Children With High-Functioning Autism Spectrum Disorders and Anxiety
Brief Title: Treatment for Children With Autism and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 03-0245
Record Dates: First submitted 2012-10-30; First posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-10

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Facing Your Fears (Experimental): FYF is a group CBT approach to managing anxiety symptoms in children with high-functioning autism spectrum disorders and anxiety.
  Interventions: Behavioral: Facing Your Fears

INTERVENTIONS:
Behavioral: Facing Your Fears — FYF is a group cognitive behavior therapy that includes parent and child participation. Groups meet weekly for 1 1/2 hours duration, for 14 consecutive weeks.

SUMMARY:
Children with high-functioning autism spectrum disorders (ASD) are at high risk for developing significant anxiety symptoms. Cognitive behavior therapies (CBT) are frequently used for children with anxiety symptoms with good success. The purpose of the current study was to examine the efficacy of a family-focused group CBT program (Facing Your Fears [FYF]) compared to Treatment As Usual (TAU). Participants were randomized to either active treatment or TAU. It was hypothesized that children who completed the active treatment would demonstrate improvement in their anxiety symptoms relative to children in TAU.

DETAILED DESCRIPTION:
Children with ASD and anxiety in our initial studies have displayed reductions in anxiety symptoms following the delivery of the FYF intervention. Given these initial successes, there are two primary purposes of this study. First, to train outpatient clinicians to fidelity on the FYF intervention for 8-14 year old children with high-functioning ASD and clinical anxiety. Second, to develop an optimal training model for learning the FYF intervention. The primary aims of Phase 1 are to develop a training manual and deliver a workshop on the FYF model to a group of outpatient clinicians in preparation for the clinicians to deliver the FYF intervention to four groups of children with ASD and anxiety. In Phase 2, the primary aims include comparing three instruction methods of learning to clinicians at three different outpatient clinics, by assessing increases in clinicians' acquisition of the intervention techniques and estimating the degree of reduction in anxiety symptoms on the primary outcome measures for the children with ASD. Instruction methods are: a) Manual, b) Workshop, c) Workshop-Plus. We hypothesize that clinicians receiving the Workshop-Plus (workshop plus ongoing consultation) condition will achieve treatment fidelity at a faster rate than clinicians receiving the other two instruction methods, and the children with ASD in the Workshop-Plus condition will display greater reductions in anxiety symptoms compared to the children in the other two conditions.

ELIGIBILITY:
Inclusion criteria:

* Clinicians must (1) be at the level of graduate student (or higher) in either a masters or doctoral program in clinical, counseling or school psychology; and (2)be working in an outpatient clinical setting serving children with ASD
* Children must (1) be 8-14 years of age; (2) living with someone who can give informed consent to participate;
* Children must have a diagnosis of ASD as defined by (a) Autism Diagnostic Observation Schedule (ADOS; Lord et al. 1999) score above spectrum cutoff; (b) Social Communication Questionnaire (SCQ; Berument et al. 1999) score above cutoff; and (c) clinical diagnosis of an ASD as determined by a review of history and current clinical presentation by a clinical psychologist and assigning one of the following diagnoses: Autistic Disorder, Asperger's Disorder, or Pervasive Developmental Disorder - Not Otherwise Specified.
* Children must have an estimated Verbal IQ of 80 or above as determined through standardized cognitive testing using the Wechsler Abbreviated Scales of Intelligence (WASI; Wechsler, 2002), or an equivalent measure of intelligence that has been administered within the past two years, and attempts to engage verbally with the examiner during the administration of Module 3 of the ADOS.
* Children must be able to read at a mid-2nd-grade level: Many activities involve narrative approaches and early reading is a pre-requisite skill for this intervention package; (as assessed by the Letter-Word Identification and Reading Comprehension subtests of the Woodcock Johnson Achievement Tests - Third Edition; WJ-III; Woodcock, McGrew, & Mather, 2001).
* Children must evince clinically significant symptoms of either , SAD, GAD, or SP anxiety and this impairment is "primary" or more functionally significant than another disorder (such as depression) as determined by the clinician evaluator. Children with clinically significant scores on SpP will also be included, although SpP cannot be the sole anxiety diagnosis for the child.
* Parents must (1) be the parent of a child with ASD and clinical anxiety as defined above and can give consent for the child to participate in the study; and (2) include men and women between the ages of 24-65.

Exclusion Criteria:

* Clinician-trainees: (1) Inability to attend at least 11/14 group sessions
* Children: (1) child is not fluent in English; (2) family cannot commit to having a minimum of 1 parent and 1 child attending 11 of 14 sessions within the intervention period; (3) child presents with psychosis, severe aggressive behavior, or other severe clinical symptoms that require more intensive treatment such as day treatment or hospitalization; (4) family plans to seek additional psychosocial treatment for anxiety during enrollment through treatment; (5) child is not able to separate from parent for a minimum of 30 minutes within the qualifying sessions; Because the parent and child interventions occur simultaneously, if a child has significant issues separating from the parent, it makes it difficult for the parent to participate in their portion of the assessment.
* Parents: (1) Parent is not fluent in English; (2) Parent is unable to attend 11/14 sessions within the intervention period

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Global Impression Scale - Improvement and Severity (CGIS-S; CGIS-I) | Administered pre and post intervention up to 12 months after final session
  CGIS-S and CGIS-I ratings were completed by an independent clinical evaluator based on scores derived from the ADIS-P and the SCARED. They were compared pre and post treatment to monitor change in anxiety symptoms.

SECONDARY OUTCOMES:
Anxiety Disorders Interview Survey for Children-Parent Version (ADIS-P) | Administered pre and post intervention up to 12 months after the final session
  The ADIS-P is a semi-structured psychiatric interview designed to assess the presence of psychiatric diagnoses, specifically anxiety disorders. Ratings were compared pre and post intervention to monitor change in anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Judy Reaven, PhD, Principal Investigator — UC Denver